CLINICAL TRIAL: NCT05917834
Title: Comparison of Nipple-areolar Complex Sensation According to Incision Types in Nipple-sparing Mastectomy
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2019-0235
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Nipple Sparing Mastectomy
Keywords: NAC sensory; Mastectomy; NSM
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Imframammary: Imframammary- NSM using imframammary incision
  Interventions: Biological: Nipple sparing mastecomy with different incision placements
- Radial/Peri-areolar: Radial/Peri-areolar- NSM using Radial/Peri-areolar incision
  Interventions: Biological: Nipple sparing mastecomy with different incision placements

INTERVENTIONS:
Biological: Nipple sparing mastecomy with different incision placements — Nipple sparing mastectomy was performed using Radial/Peri-areolar incision or imframammary incision

SUMMARY:
This study aims to assess nipple areolar complex sensation after nipple sparing mastectomy and compare the results according to different incisional approaches; specifically, inframammary fold (IMF) versus peri-areolar/radial. One-hundred-and-five post NSM patients from Oct 2019 to Nov 2021 have been recruited prospectively and evaluated for NAC sensory. A total of 97 patients (IMF 65 and peri-areolar/radial 32) were included in the analyses for comparison during follow up from 24 to 48 months after surgery. It was hypothesized that patients with IMF would have better outcomes for NAC senroy.

ELIGIBILITY:
Inclusion Criteria:

1. Females who are older than 18
2. Patients who underwent nipple sparing mastectomy in Gangnam Severance Hospital

Exclusion Criteria:

1. Loss or excision of NAC due to post-surgical necrosis
2. Diagnosis of other conditions that may interfere with cutaneous sensation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer undergoing nipple sparing mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Loss of NAC sensory by pinprick test | 2-4 years after surgery
  Difference in NAC sensory loss between the patients with two different incisions.

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea